CLINICAL TRIAL: NCT05068635
Title: Evaluation of the Efficacy of Distal Gastrectomy for the Treatment of Gastric Cancer (a Case Series)
Status: Completed | Type: Observational
Sponsor: Sylvestre KABURA (Other)
Responsible Party: Sponsor-Investigator, Sylvestre KABURA, Principal investigator, Centre Hospitalier Universitaire Ibn Rochd
Organization: Centre Hospitalier Universitaire Ibn Rochd (Other)
Other Study IDs: SK2021
Record Dates: First submitted 2021-09-20; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Gastric Cancer
Keywords: gastric cancer, gastric adenocarcinoma, total gastrectomy, subtotal gastrectomy, distal gastrectomy.
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Case series of a retrospective study of patients operated for distal adenocarcinoma of the stomach, either by total gastrectomy or distal gastrectomy at Ibn Rochd University Hospital in Casablanca, with the analysis of outcome of patients on a follow up periode of three years and eight months.

DETAILED DESCRIPTION:
Thirty (30) patients were treated for gastric cancer and were included in this study. The average age was 64 years, the sex ratio 1.5. Twenty eight patients underwent a distal gastrectomy and 2 patients underwent total gastrectomy. The median number of lymph nodes resected was 6 following distal gastrectomy versus 26 after total gastrectomy. Resection margins were clean except for three patients who underwent a distal gastrectomy. Postoperative complicationsoccured in 05 patients. They were mainly infectious, anastomotic leakage. Two 2 cases of postoperative mortality (<30 days) among patients with distal gastrectomy was noted. A progression to metastasis was found in 3 patients with subtotal gastrectomy, two of whom had insufficient lymph node clearance, compared to no cases of metastasis in patients with total gastrectomy.

ELIGIBILITY:
Inclusion Criteria: Patients bwith gastric cancer with histologic confirmation

Exclusion Criteria: Incomplete patients records

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study concerns patients who have been treated in our service for gastric cancer from fifteen years to unlimited age
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Number of patients who died for gastric cancer after distal gastrectomy | Fourty four months
  Mortality rate for patients who underwent distal gastrectomy for gastric cancer
Number of patients who developped morbidity after subgastrectmy for gastric cancer | Forty for months
  Mortality rate for patients who underwent distal gastrectomy for gastric cancer

IPD SHARING:
Plan to Share IPD: Undecided